CLINICAL TRIAL: NCT00610363
Title: A Multi-Center, Randomized, Double-Blind, Placebo Controlled Study, Tolerability, and Efficacy of Rilonacept for the Prevention of Gout Flares During Initiation of Allopurinol Therapy
Brief Title: Study of the Safety and Effectiveness of Rilonacept for the Prevention of Gout Flares
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IL1T-GA-0619
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — rilonacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Two subcutaneous injections of Placebo (for Rilonacept) as a loading dose on Day 1 followed by a single injection once a week (qw) from Week 1 to Week 16.
  Interventions: Other: Placebo (for Rilonacept)
- Rilonacept 160 mg (Experimental): Two subcutaneous injections of Rilonacept 160 mg (for a total of 320 mg) as a loading dose on Day 1, followed by a single 160 mg injection of Rilonacept qw from Week 1 to Week 16.
  Interventions: Biological: Rilonacept

INTERVENTIONS:
Biological: Rilonacept — Rilonacept 320 mg loading dose on Day 1 followed by Rilonacept 160 mg/2 mL injections qw for 17 weeks.
  Arms: Rilonacept 160 mg
Other: Placebo (for Rilonacept) — Placebo loading dose on Day 1 followed by single placebo injections (2 mL) qw for 17 weeks.
  Arms: Placebo

SUMMARY:
This was a clinical research study to determine the safety and effectiveness of an experimental drug called rilonacept in participants with gout who were beginning another additional treatment. Participants participated in this study for approximately 24 weeks. Rilonacept was being studied for use in preventing gout attacks in participants who had gout.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than 18 years of age;
* Previously met the preliminary criteria of the American Rheumatism Association (ARA) for the classification of the acute arthritis of primary gout;
* At least 2 gout flares in the year prior to the screening visit.

Exclusion Criteria:

* Acute gout flare within 2 weeks of the screening visit and during screening;
* Persistent chronic or active infections;
* History of an allergic reaction to allopurinol;
* History or presence of cancer within 5 years of the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirletta King-Davis, Study Director — Regeneron Pharmaceuticals
Locations (33):
- United States (33):
  - San Diego, California
  - Santa Maria, California
  - Whittier, California
  - Colorado Srings, Colorado
  - DeLand, Florida
  - Ocala, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Dunwoody, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Indianapolis, Indiana
  - South Bend, Indiana
  - Owensboro, Kentucky
  - Wheaton, Maryland
  - Billings, Montana
  - Omaha, Nebraska
  - Reno, Nevada
  - Albany, New York
  - Plainview, New York
  - Roslyn, New York
  - Monroe, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Mayfield Village, Ohio
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - West Reading, Pennsylvania
  - Charleston, South Carolina
  - Grenville, South Carolina
  - Dallas, Texas
  - Spokane, Washington

REFERENCES:
- [Derived] Schumacher HR Jr, Sundy JS, Terkeltaub R, Knapp HR, Mellis SJ, Stahl N, Yancopoulos GD, Soo Y, King-Davis S, Weinstein SP, Radin AR; 0619 Study Group. Rilonacept (interleukin-1 trap) in the prevention of acute gout flares during initiation of urate-lowering therapy: results of a phase II randomized, double-blind, placebo-controlled trial. Arthritis Rheum. 2012 Mar;64(3):876-84. doi: 10.1002/art.33412. PMID 22223180
- [Derived] Khanna D, Sarkin AJ, Khanna PP, Shieh MM, Kavanaugh AF, Terkeltaub RA, Lee SJ, Singh JA, Hirsch JD. Minimally important differences of the gout impact scale in a randomized controlled trial. Rheumatology (Oxford). 2011 Jul;50(7):1331-6. doi: 10.1093/rheumatology/ker023. Epub 2011 Mar 3. PMID 21372003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 27 study sites in United States (US) between 19 November 2007 and 16 October 2008. A total of 154 participants were screened in the study.
Pre-assignment Details: Out of 154 participants, 83 were randomized and treated in the study. Participants were randomized in 1:1 ratio to receive either Placebo or Rilonacept 160 mg.
Period: Overall Study
Arm/Group | Placebo | Rilonacept 160 mg
Started | 42 | 41
Completed | 31 | 38
Not Completed | 11 | 3
Not completed — Non-compliance with protocol | 0 | 1
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other than specified above | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline population included full analysis set (FAS) comprising of all randomized participants who received any study medication and was based on treatment allocated by Interactive voice response system (IVRS) at randomization (as randomized).
Groups:
- Placebo: Two subcutaneous injections of Placebo (for Rilonacept) as a loading dose on Day 1 followed by a single injection qw from Week 1 to Week 16.
- Total: Total of all reporting groups
Arm/Group | Placebo | Rilonacept 160 mg | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11.59) | 51.9 (10.61) | 51.0 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 40 | 40 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 41 | 40 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 3 | 2 | 5
  White | 38 | 36 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Gout Flares Per Participant Assessed From Day 1 to Day 84 (Week 12)
Description: A gout flare was defined as participant reported acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Number of gout flares per participant was reported for this outcome measure. For drop-outs, only flares occurred before Day 84 were counted, regardless whether the flares occurred during the treatment period or not.
Time Frame: Day 1 (Baseline) to Day 84 (Week 12)
Population: Full analysis set (FAS) that included all randomized participants who received any study medication and was based on treatment allocated by IVRS at randomization (as randomized).
Measure: Mean (Standard Deviation); unit: Number of gout flares per participant
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 42 | 41
Number of gout flares per participant | 0.79 (1.071) | 0.15 (0.358)

2. Secondary Outcome: Percentage of Participants With at Least One Gout Flare From Day 1 to Day 84 (Week 12)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain; and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Percentage of participants with at least one gout flare was reported for this outcome measure.
Time Frame: Day 1 (Baseline) to Day 84 (Week 12)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 42 | 41
percentage of participants | 45.2 | 14.6

3. Secondary Outcome: Mean Number of Gout Flares Per Month Per Participant From Day 1 to Day 84 (Week 12)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain, and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Mean number of flares per month = (total number of flares observed)/ (total number of days subject was in the period/28 days).
Time Frame: Day 1 (Baseline) to Day 84 (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of gout flares
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 42 | 41
number of gout flares | 0.30 (0.424) | 0.06 (0.178)

4. Secondary Outcome: Mean Number of Gout Flare Days Per Participant From Day 1 to Day 84 (Week 12)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain, and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Mean number of gout flare days per participant was reported for this outcome measure.
Time Frame: Day 1 (Baseline) to Day 84 (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Gout flare days
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 42 | 41
Gout flare days | 5.17 (8.015) | 1.41 (5.230)

5. Secondary Outcome: Mean Number of Gout Flare Days Per Month Per Participant From Day 1 to Day 84 (Week 12)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain, and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Mean number of gout flare days per month per participant was reported for this outcome measure.
Time Frame: Day 1 (Baseline) to Day 84 (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Gout flare days
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 42 | 41
Gout flare days | 2.09 (3.608) | 0.52 (1.779)

6. Secondary Outcome: Number of Gout Flare Days With Participant's Pain Score of 5 or More (From Daily Diary) Per Participant From Day 1 to Day 84 (Week 12)
Description: Participants were asked to complete a telephone diary by calling the IVRS daily beginning at the baseline visit (Day 1) through the follow-up visit (Day 154) and reported their general well-being, gout symptoms, and weekly study drug administrations. At the onset of pain from a gout flare, participants were to answer additional diary questions regarding their gout flare and had to continue daily flare assessments until they reported the flare had ended. If a flare occurred just prior to the follow-up visit (Day 154), participants were to continue completing the daily diary until the flare resolved. Gout flare pain was assessed on a scale from 0 to 10 (with 0=no pain and 10=severe pain) within the past 24 hours.
Time Frame: Day 1 (Baseline) to Day 84 (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Gout flare days
Groups:
- Placebo: Two subcutaneous injections of Placebo (for Rilonacept ) as a loading dose on Day 1 followed by a single injection qw from Week 1 to Week 16.
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 42 | 41
Gout flare days | 2.02 (4.51) | 0.22 (0.79)

7. Secondary Outcome: Number of Gout Flare Days With Participant's Pain Score of 5 or More (From Daily Diary) Per Month Per Participant From Day 1 to Day 84 (Week 12)
Description: Participants were asked to complete a telephone diary by calling the IVRS daily beginning at the baseline visit (Day 1) through the follow-up visit (Day 141) and reported their general well-being, gout symptoms, and weekly study drug administrations. At the onset of pain from a gout flare, participants were to answer additional diary questions regarding their gout flare and had to continue daily flare assessments until they reported the flare had ended. If a flare occurred just prior to the follow-up visit (Day 141), participants were to continue completing the daily diary until the flare resolved. Gout flare pain was assessed on a scale from 0 to 10 (with 0=no pain and 10=severe pain) within the past 24 hours.
Time Frame: Day 1 (Baseline) to Day 84 (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Gout flare days
Arm/Group | Placebo | Rilonacept 160 mg
Number analyzed (Participants) | 42 | 41
Gout flare days | 0.87 (2.05) | 0.07 (0.26)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 22) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that developed/worsened during the 'on treatment period' (time from the administration of first dose of study drug through the period ending 42 days after the last dose of study drug). Analysis was performed on safety population the included all participants who received any study medication and were analyzed according to the treatment actually received (as treated).
Arm/Group | Placebo | Rilonacept 160 mg
Serious Adverse Events (participants affected / at risk) | 2/42 | 1/41
Other Adverse Events (participants affected / at risk) | 8/42 | 6/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | Rilonacept 160 mg (N=41)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | Rilonacept 160 mg (N=41)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Gout (Metabolism and nutrition disorders) | 3 (7) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI/Institution will provide a copy of any publication to Sponsor prior to submission for review. Sponsor may request to remove confidential information from submission, provided that removal does not preclude the complete and accurate presentation and interpretation of the study results.